CLINICAL TRIAL: NCT03719495
Title: Evaluation of the Effects of Endocrine Therapies on Immune Cell Repertoire and Function in Early Stage Estrogen Receptor Positive Breast Cancer Patients
Brief Title: Evaluation of Endocrine Therapy Effects of Host Immunity in Early Stage Breast Cancer
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: Pro00100408
Record Dates: First submitted 2018-10-15; First posted 2018-10-25 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; Estrogen Receptor-positive Breast Cancer; Healthy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and archival tumor tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cohort 1: Pre-menopausal women as healthy controls will be recruited on Duke University Campus and Duke University Hospital.
- Cohort 2: Postmenopausal women as healthy controls will be recruited on Duke University Campus and Duke University Hospital.
- Cohort 3: Pre-menopausal women initiating tamoxifen after standard of care local-regional therapy after surgery +/- radiation.
- Cohort 4: Pre-menopausal women initiating ovarian suppression plus aromatase inhibition after surgery +/- radiation.
- Cohort 5: Postmenopausal women initiating endocrine therapy with aromatase inhibition after standard of care surgery +/- radiation.

SUMMARY:
The purpose of this research study is to learn about the effects that standard of care endocrine therapies have on the immune system's response to cancer by looking at the number and types of immune cells present and how they function in women with early stage estrogen receptor positive (ER+) breast cancer.

DETAILED DESCRIPTION:
The study will enroll mainly subjects with estrogen receptor positive breast cancer that have completed surgery and radiation therapy to remove the tumor(s) and have not yet started standard treatment endocrine therapy. There is one group of subjects who have not been diagnosed with cancer. The information learned from this study will help doctors understand more about how the immune system responds to endocrine therapy for early stage breast cancer in people who are estrogen receptor positive with the goal of developing improved therapies that harness the immune system.

ELIGIBILITY:
Inclusion Criteria health cohorts:

1. No known significant health problems.
2. Available to participate for the planned duration of the investigational study (6 months).
3. Able and willing to complete the informed consent process.
4. Agree to have blood stored for future studies.
5. Premenopausal women must have a history of regular menses defined as occuring monthly at regular intervals.
6. Postmenopausal women are defined as:

   * prior bilateral oophorectomy
   * 60 or older
   * age less than 60 years

     * amenorrheic for 12 months or more in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression
     * and follicle-stimulating hormone (FSH) and plasma estradiol in the postmenopausal range.

Inclusion Criteria (All endocrine therapy cohorts):

1. Early stage breast cancer including T1-3, N0-3.
2. Histologically documented estrogen receptor positive adenocarcinoma of the breast that is (any progesterone status allowed):

   * ER positive defined as ≥ 10% tumor cells positive for ER by immunohistochemistry (IHC), irrespective of staining intensity.
   * HER2 negative status is determined by:

     * IHC 1+, as defined by incomplete membrane staining that is faint/barely perceptible and within >10% of invasive tumor cells, OR
     * IHC 0, as defined by no staining observed or membrane staining that is incomplete and is faint/barely perceptible and within ≤ 10% of the invasive tumor cells, OR
     * FISH negative based on:

       * Single-probe average HEr2 copy number <4.0 signals/cell, OR
       * Dual-probe HER2/CEP17 ratio <2.0 with an average HER2 copy number <4.0 signals/cell.
3. Patients should have plans to initiate standard of care endocrine therapy in the adjuvant setting per primary provider.
4. Patients can have had neoadjuvant or adjuvant chemotherapy with resolution of all hematologic toxicity to less than grade 1 by CTCAE v4.0 (e.g. Hg ≥10d/dL, Platelets 75,000mm3, Neutrophil >1500mm3).
5. Patients should be willing to provide an archival tumor specimen from their definitive surgery.
6. Able and willing to complete the informed consent process.
7. Available to participate for the planned duration of the study (6 months).
8. Agree to have bio-specimens stored for future research.

Exclusion Criteria (all cohorts):

1. Relapsed or metastatic breast cancer.
2. History of cancer or concurrent active malignancy (excluding basal cell skin cancer, resected squamous cell carcinoma of the skin).
3. Receipt of neoadjuvant or previous endocrine therapy including ovarian function suppression in the neoadjuvant setting.
4. Current use of hormonal birth control (copper IUD allowed) or estrogen replacement therapy.
5. Known to have a condition in which repeated blood draws pose more than minimal risk for the subject such as hemophilia, other severe coagulation disorders or significantly impaired venous access.
6. Concurrent enrollment in a therapeutic clinical trial involving novel drug therapies
7. Active autoimmune disease that has required systemic treatment in past year (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, or similar treatment) is not considered a form of systemic treatment.
8. Immunodeficient subjects, E.G., receiving systemic steroid therapy or any other form of immunosuppressive therapy within 30 days prior to the first dose of endocrine therapy treatment
9. Concurrent use of other oncologic therapies in the adjuvant setting other than bisphosphonates
10. Active or ongoing infection
11. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease, active bleeding diatheses including any subjects known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness / social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
12. Pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pre-menopausal and postmenopausal women with breast cancer who are initiating endocrine therapy or aromatase inhibitors.
  Pre-menopausal and postmenopausal healthy women who are not on any hormonal birth control.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Changes in estrogen levels in response to adjuvant endocrine therapy. | 2 years
  Phenotypic and functional characterization of T cell and B cell populations will be performed on peripheral blood mononuclear cells.

SECONDARY OUTCOMES:
Changes in regulatory T cells in premenopausal vs postmenopausal women treated with aromatase inhibitors. | Through study completion, approximately 1 year.
  Blood will be assessed at each time point to understand the impact of endocrine therapy on regulatory T cells.
Changes in T cell activation/ V cell activation in premenopausal vs postmenopausal women treated with aromatase inhibitors. | Through study completion, approximately 1 year.
  Blood will be assessed at each time point to understand the impact of endocrine therapy in T cell activation/ V cell activation.
Changes in T cell exhaustion in premenopausal vs postmenopausal women treated with aromatase inhibitors. | Through study completion, approximately 1 year.
  Blood will be assessed at each time point to understand the impact of endocrine therapy in T cell exhaustion.
Changes in myeloid-derived suppressor cells in premenopausal vs postmenopausal women treated with aromatase inhibitors. | Through study completion, approximately 1 year.
  Blood will be assess at each time point to understand the impact of endocrine therapy on myeloid-derived suppressor cells.
Changes in physical manifestations with the Patient-Reported Outcomes Measurement Information System (PROMIS) fatigue survey to measure response to adjuvant endocrine therapy. | Through study completion, approximately 1 year.
  PROMIS Fatigue quality of life survey will be given at each time point.
Changes in inflammatory markers with Patient-Reported Arthralgia Inventory (PRAI) to measure response to adjuvant endocrine therapy. | Through study completion, approximately 1 year.
  16-item Patient-Reported Arthralgia Inventory (PRAI) quality of life survey will be given at each time point.
Assess changes in RNA express in response to endocrine therapy. | Through study completion, approximately 1 year.
  RNA expression of PMBCs will be performed to assess changes in gene expression due to endocrine therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Dent, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States